CLINICAL TRIAL: NCT01785251
Title: Haemodynamic Performance of Neuromuscular Electrical Stimulation (NMES) During Recovery From Total Hip Arthroplasty
Brief Title: Neuromuscular Electrical Stimulation Following Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Irish Research Council (Other); Mid Western Regional Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Gearoid O Laighin, Professor, National University of Ireland, Galway, Ireland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EE-NMES-DVT-011
Record Dates: First submitted 2013-02-01; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Deep Vein Thrombosis; Total Hip Arthroplasty
Keywords: Neuromuscular electrical stimulation; NMES; Deep vein thrombosis; DVT; total hip arthroplasty; lower limb hemodynamics
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NMES (Experimental): Application of neuromuscular electrical stimulation to the calf muscles of the patient in order to elicit contraction of the calf muscle pump and thus, eject venous blood proximally.
  Interventions: Device: Neuromuscular Electrical Stimulation

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation — Applied using a custom built, medically approved stimulator called the Duo-STIM. NMES to be applied to the calf muscles to elicit a muscular contraction to eject blood through the venous system.

SUMMARY:
Patients post total hip arthroplasty (THA) remain at high risk of developing Deep Vein Thrombosis (DVT) during the recovery period following surgery despite the availability of effective pharmacological and mechanical prophylactic methods. The use of calf muscle neuromuscular electrical stimulation (NMES) during the hospitalised recovery period on this patient group may be effective at preventing DVT. However, the haemodynamic effectiveness and comfort characteristics of NMES in post-THA patients immediately following surgery have yet to be established.

The main objectives are:

1. To establish if patients in the early post-operative period have tolerance for NMES.
2. To determine if applying NMES to patients immediately post-THA increases venous outflow from the lower limb over resting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent total hip arthroplasty the previous day

Exclusion Criteria:

* Patients with Diabetes Mellitus
* Patients with Peripheral Vascular Disease
* Patients currently involved in another trial
* Previous diagnosis of DVT

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Lower limb haemodynamic performance | 4 hours
  Duplex Doppler ultrasound will be used as the outcome measure. Both legs will be measured for hemodynamic performance in the popliteal vein by placing the probe at the popliteal fossa.
  Measurements of peak venous velocity (cm/s), popliteal vein diameter (cm), time averaged mean velocity (TAMEAN, cm/s) and volume flow (ml/min) will be recorded.
  Doppler measurements will be taken initially at rest, before the application of NMES and once again when the NMES session had commenced.

SECONDARY OUTCOMES:
Patient comfort during application of NMES | 4 hours
  Measurements will be taken at 3 time points (before application of NMES, after application of NMES had begun and at the end of the protocol).
  The measurement consists of asking patients to mark their level of comfort using a 100mm, non-hatched visual-analogue-scale (VAS).
  A VAS of 30 mm or less will be categorised as mild pain, between 31 and 69mm as moderate pain and scores of 70mm or greater as severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Gearóid ÓLaighin, BEng, MEng, PhD, Principal Investigator — National University of Ireland, Galway
Locations (1):
- Mid-Western Regional Orthoapedic Hospital Croom, Limerick, Ireland

REFERENCES:
- [Derived] Broderick BJ, Breathnach O, Condon F, Masterson E, Olaighin G. Haemodynamic performance of neuromuscular electrical stimulation (NMES) during recovery from total hip arthroplasty. J Orthop Surg Res. 2013 Mar 5;8:3. doi: 10.1186/1749-799X-8-3. PMID 23497524